CLINICAL TRIAL: NCT04314687
Title: Allogeneic Umbilical Cord Mesenchymal Stem Cells and Conditioned Medium for Cerebral Palsy in Children
Brief Title: Stem Cell and Conditioned Medium for Cerebral Palsy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PT. Prodia Stem Cell Indonesia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: CT/CP/02/2020
Record Dates: First submitted 2020-02-20; First posted 2020-03-19 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Cerebral Palsy
Keywords: Allogeneic Mesenchymal Stem Cells; Umbilical Cord Mesenchymal Stem Cells; Intrathecal Injection; Cerebral Palsy; Conditioned Medium
MeSH Terms: conditions — Cerebral Palsy | interventions — Culture Media, Conditioned; Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- UCMSCs + CM (Experimental): UCMSCs + CM is administered via intrathecal injection
  Interventions: Biological: Umbilical Cord Mesenchymal Stem Cells; Biological: Conditioned Medium
- UCMSCs (Experimental): UCMSCs is administered via intrathecal injection
  Interventions: Biological: Umbilical Cord Mesenchymal Stem Cells
- Standard Therapy (Active Comparator): Physiotherapy
  Interventions: Other: Standard Therapy

INTERVENTIONS:
Biological: Umbilical Cord Mesenchymal Stem Cells — The umbilical cord was removed from the donor and brought to cell culture facility immediately. Upon arrival, pre-sterility sample testing was performed to ensure the sample was free from contaminant. Culture processes were conducted in a laboratory room where high sterility and safety were guaranteed. Every batch of the cells was monitored by a series of quality control testing to assure the quality of the product.
  Other Names: Allogeneic Mesenchymal Stem Cells
  Arms: UCMSCs; UCMSCs + CM
Biological: Conditioned Medium — Conditioned medium collected from umbilical cord mesenchymal stem cell (UC-MSC) cultured. Every batch of the conditioned medium was monitored by a series of quality control testing to assure the quality of the product.
  Other Names: Umbilical Cord Mesenchymal Stem Cells derived Conditioned Medium
  Arms: UCMSCs + CM
Other: Standard Therapy — Standard therapy for cerebral palsy such as physiotherapy
  Other Names: Physiotheraphy
  Arms: Standard Therapy

SUMMARY:
The aim of this study was to compare the effectiveness of umbilical cord mesenchymal stem cells (UCMSCs) and conditioned medium (CM) administration, UCMSCs only and control with standard therapy.

Hypothesis: UCMSCs + CM therapy resulting in higher improvement in cognitive function, gross motor function and chemical factors than UCMSCs and standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as Cerebral palsy with total body involvement type
* Age between 6 month - 3 years old
* Parents requesting for cell therapy
* The parents give sign in informed consent form do to examination, therapy, blood sampling collection and observation for their child

Exclusion Criteria:

* Head circumference less than -3 SD (more than 3 cm) Nellhaus standard
* Have diagnosed meningitis and encephalitis
* Have diagnosed congenital infection i.e. toxoplasmosis, rubella congenital, cytomegalovirus
* Have diagnosed metabolic disorder, chromosome disorder, congenital malformation or neuroregeneratif disease
* Progressive disorder
* Regressive development disorder
* Severe anatomical abnormalities in Brain MRI

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2023-09-25 (Estimated); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function | 3 month after stem cells
  Gross Motor Function Classification System (GMFCS)
Gross Motor Function | 6 month after stem cells
  Gross Motor Function Classification System (GMFCS)
Gross Motor Function | 3 month after stem cells
  Gross Motor Function Measure (GMFM)
Gross Motor Function | 6 month after stem cells
  Gross Motor Function Measure (GMFM)
Cognitive Function | 3 month after stem cells
  Bayley Scales of Infant Development (BSID) version III
Cognitive Function | 6 month after stem cells
  Bayley Scales of Infant Development (BSID) version III

SECONDARY OUTCOMES:
Chemical Marker | 3 month after stem cells
  Insulin-like growth factor 1 (IGF-1); stromal derived factor-1α (SDF-1α); brain derived neurotrophic factors (BDNF), Vascular endothelial growth factor (VEGF),glial cell line-derived neutrophic factor (GDNF), fibroblast growth factor (FGF), Doublecortin (DCX)
Chemical Marker | 6 month after stem cells
  Insulin-like growth factor 1 (IGF-1); stromal derived factor-1α (SDF-1α); brain derived neurotrophic factors (BDNF), Vascular endothelial growth factor (VEGF),glial cell line-derived neutrophic factor (GDNF), fibroblast growth factor (FGF), Doublecortin (DCX)

CONTACTS AND LOCATIONS:
Locations (1):
- Indonesian National Brain Center, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No